CLINICAL TRIAL: NCT01823289
Title: Clinical Efficacy and Safety of Itraconazole Injection/Oral Solution Sequential Therapy for Treatment of Invasive Pulmonary Fungal Infections
Brief Title: An Efficacy and Safety Study of Itraconazole Sequential Therapy (Intravenous Injection Followed by Oral Solution) in Invasive Pulmonary Fungal Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014362; ITRFUN4025; SPOIV-CHN-MA-04
Record Dates: First submitted 2013-03-12; First posted 2013-04-04 (Estimated); Results first posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-04

CONDITIONS: Pulmonary Fungal Infection
Keywords: Invasive Pulmonary Fungal Infection; Itraconazole
MeSH Terms: conditions — Lung Diseases, Fungal | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Itraconazole Sequential Therapy (Experimental)
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Itraconazole — Itraconazole 200 milligram (mg) intravenous injection will be given twice daily for first 2 days, 200 mg once daily for the subsequent 12 days, then sequential itraconazole oral solution 200 mg twice daily will be given for 2 to 4 weeks.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of itraconazole sequential therapy (intravenous injection/oral solution) in participants with invasive pulmonary fungal infections ([IPFI]; lung diseases caused by fungal infection).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single arm, multicenter (when more than one hospital or medical school team work on a medical research study) study to evaluate the efficacy and safety of itraconazole sequential therapy in participants with IPFI. The study duration will be 4 to 6 weeks. The treatment will be divided into the intravenous (into a vein) injection period and the oral solution administration (giving) period. During the intravenous injection period 200 milligram (mg) twice daily loading dose (large initial dose) will be given for first 2 days, 200 mg once daily for the subsequent 12 days. Then sequential itraconazole oral solution 200 mg twice daily will be given as maintenance therapy (treatment designed to help the original primary treatment to succeed) for 2-4 weeks. Participant's clinical, mycological and comprehensive efficacy will be assessed at Week 6. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Probable or proven invasive pulmonary infectious participants (IPFI) - Hospitalized participants (at least hospitalized treatment and observation could be ensured during the intravenous injection period) - The participants (or legal representatives) have signed the informed consent forms.

Exclusion Criteria:

* Currently taking taboo drugs, such as terfenadine, astemizole, cisapride and HMG CoA reductase inhibitors (for example simvastatin, lovastatin, oral or intravenous midazolam or triazolam) - History of allergy or intolerance to imidazoles or pyrrole drugs (for example fluconazole, itraconazole, ketoconazole, miconazole, clotrimazole) - Pregnant and breast feeding women, or women of child bearing age not taking effective contraception measures - Participants with pure oral, urinary tract, and vaginal candidiasis (yeast infection) - Participants with fungal meningitis (inflammation of the meninges), active liver disease, renal insufficiency with the serum creatinine clearance rate less than 30 milliliter per minute (ml/min), and current abnormal cardiac function such as congestive heart failure (condition in which the heart is unable to pump out sufficient blood to meet the metabolic need of the body), or participants with history of congestive heart failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-06; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical trial, Study Director — Xian-Janssen Pharmaceutical Ltd.

RESULTS

PARTICIPANT FLOW:
Groups:
- Itraconazole Sequential Therapy: Itraconazole 200 milligram (mg) intravenous (directly into the vein) injection was given twice daily for first 2 days and once daily for the subsequent 12 days, then sequential itraconazole oral solution 200 mg twice daily was given for 2 to 4 weeks.
Period: Overall Study
Arm/Group | Itraconazole Sequential Therapy
Started | 71
Completed | 47
Not Completed | 24
Not completed — Lost to Follow-up | 5
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 1
Not completed — Physician Decision | 9
Not completed — Administered contraindicated medicine | 1
Not completed — Transaminase increased more than 3 times | 1
Not completed — Drug affected efficacy and safety | 1
Not completed — Creatinine clearance<30milliliter/minute | 1

BASELINE CHARACTERISTICS:
Arm/Group | Itraconazole Sequential Therapy
Number analyzed (Participants) | 60
Age Continuous [Median (Full Range); unit: years] — Out of 71 total participants, baseline characteristic (age) was available for only 60 participants who were included in the full analysis set (FAS) population.
  years | 55.5 [33.34 to 79.45]
Sex: Female, Male [Count of Participants; unit: Participants] — Out of 71 total participants, baseline characteristic (gender) was available for only 60 participants who were included in the full analysis set (FAS) population.
  Participants
    Female | 23
    Male | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Efficacy
Description: Clinical efficacy was assessed as cured: the signs and symptoms of invasive fungal infections (IFI) completely disappeared or full or nearby resolution of radiographic manifestations; markedly improved: the signs and symptoms of IFI were improved or disappeared and at least 50 percent improvement of radiographic findings; improved: the signs and symptoms of IFI were moderately improved and less than 50 percent improvement of radiographic findings; failed: the clinical symptoms and signs of IFI were not changed or worsened.
Time Frame: Week 6
Population: The Full analysis set (FAS) population included all participants who received at least 1 intravenous infusion or oral solution of the study drug and completed at least 1 post-baseline visit.
Measure: Number; unit: participants
Arm/Group | Itraconazole Sequential Therapy
Number analyzed (Participants) | 60
participants
  Cured | 8
  Markedly Improved | 29
  Improved | 18
  Failed | 5

2. Primary Outcome: Number of Participants With Mycological Efficacy
Description: Mycological efficacy was assessed as fungi cleared: negative for fungal microscopic examination and culture (test for infection or organisms that could cause infection); fungi not cleared: positive for fungal microscopic examinations and/or culture.
Time Frame: Week 6
Population: The Full analysis set (FAS) population included all participants who received at least 1 intravenous infusion or oral solution of the study drug and completed at least 1 post-baseline visit. Here 'N' signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Itraconazole Sequential Therapy
Number analyzed (Participants) | 30
participants
  Fungi cleared | 20
  Fungi not cleared | 10

3. Primary Outcome: Number of Participants With Comprehensive Efficacy
Description: Comprehensive efficacy was assessed as cured: the symptoms, signs, laboratory examination and pathogenic examination were return to normal; markedly improved: the disease condition was markedly improved but symptoms, signs, laboratory examination and pathogenic examination were not return to normal; improved: the disease condition was improved to some extent after drug administration, but the improvement was not significant enough; failed: the disease condition was not improved significantly or worsened after drug administration.
Time Frame: Week 6
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Itraconazole Sequential Therapy
Number analyzed (Participants) | 60
participants
  Cured | 8
  Markedly Improved | 32
  Improved | 16
  Failed | 4

ADVERSE EVENTS:
Time Frame: From the signing of informed consent until end of the study (week 6).
Description: Safety set (SS) population (N=61) included all participants who received at least 1 dose of study drug and had safety documents.
Arm/Group | Itraconazole Sequential Therapy
Serious Adverse Events (participants affected / at risk) | 4/61
Other Adverse Events (participants affected / at risk) | 13/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Itraconazole Sequential Therapy (N=61)
Edema (General disorders) | 1
Death (General disorders) | 2
Fungal infection (Immune system disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Itraconazole Sequential Therapy (N=61)
Granulocytopenia (Blood and lymphatic system disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hyperbilirubinemia (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 3
GPT increased (Hepatobiliary disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 1
Renal function abnormal (Renal and urinary disorders) | 1
Dermatoses (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Night sweating (General disorders) | 1
Fever (General disorders) | 1
Abdominal pain (General disorders) | 1
Septic shock (General disorders) | 1
Headache (General disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Non-specific anorexia (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Palpitation (Cardiac disorders) | 1
Dizziness (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less